CLINICAL TRIAL: NCT00710996
Title: Blue Light Intraocular Lenses (IOLs) and Photostress
Status: Completed | Type: Observational
Sponsor: Alcon Research (Industry)
Responsible Party: Rick Potvin, Alcon Laboratories, Inc.
Other Study IDs: M07-023
Record Dates: First submitted 2008-07-03; First posted 2008-07-08 (Estimated); Results first posted 2010-01-29 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-01

CONDITIONS: Cataract
Keywords: AcrySof IQ IOL
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- AcrySof Natural Intraocular Lens: AcrySof Natural Intraocular Lens (IOL) - Patients with previous bilateral implant of any Alcon lens model starting with the letters "SN"
- AcrySof clear intraocular lens: AcrySof clear intraocular lens (IOL) - Patients with previous bilateral implant of any Alcon lens model starting with the letters "SA"
- Phakic patients: Phakic patients - Age matched patients who have not had cataract surgery

SUMMARY:
To determine what effect a blue light filtering Intraocular Lens (IOL) has on macular pigment levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients with existing bilateral IOLs of given type, age-matched patients with normal vision and no cataract surgery.

Exclusion Criteria:

* Age related

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with existing bilateral Intraocular Lenses (IOLs) of given type, age-matched patients with normal vision and no cataract surgery.
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2008-01; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Call Alcon Call Center for Study Locations, Fort Worth, Texas, United States

REFERENCES:
- [Derived] Hammond BR, Bernstein B, Dong J. The Effect of the AcrySof natural lens on glare disability and photostress. Am J Ophthalmol. 2009 Aug;148(2):272-276.e2. doi: 10.1016/j.ajo.2009.03.014. Epub 2009 May 7. PMID 19426959

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with existing bilateral intraocular lenses (IOLs) of given type, age-matched patients with normal vision and no cataract surgery.
Pre-assignment Details: Subjects eligibility was determined at the preoperative visit. All subjects met inclusion/exclusion criteria.
Period: Overall Study
Arm/Group | AcrySof Natural Intraocular Lens | AcrySof Clear Intraocular Lens | Phakic Patients
Started | 17 | 20 | 21
Completed | 16 | 16 | 21
Not Completed | 1 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AcrySof Natural Intraocular Lens | AcrySof Clear Intraocular Lens | Phakic Patients | Total
Number analyzed (Participants) | 17 | 20 | 21 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 3 | 7
  >=65 years | 15 | 18 | 18 | 51
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 10 | 34
  Male | 6 | 7 | 11 | 24

OUTCOME MEASURES:

1. Primary Outcome: Photostress Recovery Time in Seconds.
Description: The time necessary to recover function (e.g., contrast discrimination) following exposure to a bright glare source.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | AcrySof Natural Intraocular Lens | AcrySof Clear Intraocular Lens | Phakic Patients
Number analyzed (Participants) | 16 | 16 | 21
seconds | 36 (25.94) | 41.46 (25.94) | 24.88 (15.45)

ADVERSE EVENTS:
Time Frame: N/A - Not collected
Description: Serious and/or other [non-serious] adverse events were not collected/assessed
Arm/Group | AcrySof Natural Intraocular Lens | AcrySof Clear Intraocular Lens | Phakic Patients
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No paper that incorporates Sponsor Condfidential information will be submitted for publication without Sponsor's prior written agreement.